CLINICAL TRIAL: NCT05164029
Title: The Clinical Cohort Study of Reproductive Health
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Principal Investigator, Dan Zhang, Vice president, Women's Hospital School Of Medicine Zhejiang University
Other Study IDs: CSRH
Record Dates: First submitted 2021-12-09; First posted 2021-12-20 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Fertility Disorders; Assisted Reproductive Technology; Offspring Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ART couples: Couples in reproductive age undergoing ART treatment
  Interventions: Other: Completion questionnaires/providing biological samples
- natural pregnancy couples: Couples who get pregnant naturally
  Interventions: Other: Completion questionnaires/providing biological samples

INTERVENTIONS:
Other: Completion questionnaires/providing biological samples — Participant completes baseline interview at enrollment, then completes questionnaires and provides biological samples at each scheduled study visit.

SUMMARY:
The study will conduct a multicenter prospective clinical cohort study to collect comprehensive health information and essential specimens from pre-pregnancy to postpartum offspring development. We will combine the reproductive medicine with the big data technologies and cloud computing to explore the key factors which will induce the occurrence the reproductive disorders and effect the health of women and offspring. Based on the discovery of the cohort study, we will construct a prediction model for improvement of ART，optimizing the effectiveness and safety of ART.

DETAILED DESCRIPTION:
Safeguarding the health of women and children is an important part of The Healthy China 2030 Plan. Precisely controlling the fertility process will help to improve the quality of national population. Lots of studies have reported that environmental exposure, lifestyle, diet and other factors are related to fertility, female pregnancy and postpartum health, and offspring development. Some studies have found that assisted reproductive technology (ART) represents an increased risk of epigenetic-related diseases or birth defects.

The study will conduct a multicenter prospective clinical cohort study to collect comprehensive health information and essential specimens from pre-pregnancy to postpartum offspring development. We will combine the reproductive medicine with the big data technologies and cloud computing to explore the key factors which will induce the occurrence the reproductive disorders and effect the health of women and offspring. Based on the discovery of the cohort study, we will construct a prediction model for improvement of ART，optimizing the effectiveness and safety of ART.

ELIGIBILITY:
Inclusion Criteria:

1. Couples undergoing treatment for infertility or getting pregnant naturally and wanting to deliver their babies in study hospitals.
2. Men 22-55 years old
3. Women 20 - 45 years old

Exclusion Criteria:

1. Any individual or couple who is outside of age range .
2. Any couple who don't plan to complete their pregnancy check-up or deliver their babies in study hospitals.
3. Any couples had participated in other clinical studies.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study subjects will be recruited from couples seeking treatment of infertility or getting pregnant naturally and wanting to deliver their babies in the study hospitals. Men must be at least 22 years old and women must be at least 20 years to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
live birth rate | 1 day after delivery
  Number of women with live births / number of women randomized to the specific group.
birth weight | 1 day after delivery
  Weight of newborns at delivery.
weight | Change from the date of delivery up to 2 years after delivery
  the weight of offspring
height | Change from the date of delivery up to 2 years after delivery
  the height of offspring
Incidence of mental diseases and metabolic dysfunction | from the date of delivery up to 2 years after delivery

SECONDARY OUTCOMES:
implantation rate | 11-12 weeks after embryo transfer
  Implantation rate was defined as the percentage of fetal heart beat among total transferred embryos at 12 weeks' gestational age.
clinical pregnancy rate | 6 weeks after embryo transfer
  Clinical pregnancy was defined as an observation of gestational sac via ultrasonography.
preterm birth rate | 28 gestational weeks to 37 gestational weeks
  preterm birth is defined as gestational weeks between 28 to 37.
neonatal complication rate | 1 day after delivery
  Neonatal complication includes neonatal respiratory disorders, neonatal cerebral palsy, neonatal encephalopathy and other disease that should been sent into neonatal ICU.

IPD SHARING:
Plan to Share IPD: No
All data relevant to the study will be generated in the article or uploaded as supplementary information. Deidentified participant data will be available from Dr. Dan Zhang (zhangdan@zju.edu.cn) on a reasonable request. Protocols and statistical analysis plans will be included as supplementary information.